CLINICAL TRIAL: NCT06531538
Title: A PHASE 2, RANDOMIZED, PARTIALLY DOUBLE-BLIND TRIAL TO EVALUATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF A MULTIVALENT PNEUMOCOCCAL CONJUGATE VACCINE ADMINISTERED IN HEALTHY TODDLERS 12 THROUGH 15 MONTHS OF AGE
Brief Title: A Study to Learn About How a New Pneumococcal Vaccine Works in Children
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: C4931010; NCT06531538 (Registry Identifier: ClinicalTrials.gov); 2025-000101-16 (EudraCT Number)
Record Dates: First submitted 2024-07-23; First posted 2024-08-01 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Pneumococcal Disease
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Study is partially blinded as 2 of the 3 groups are blinded and 1 is unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- PG4 1-Dose Group (Experimental): Participants to receive a single injection of Multivalent Pneumococcal Vaccine
  Interventions: Biological: PG4
- PG4 2-Dose Group (Experimental): Participants to receive two injections of Multivalent Pneumococcal Vaccine
  Interventions: Biological: PG4
- 20-valent pneumococcal conjugate vaccine (20vPnC) (Active Comparator): Participants to receive a single injection of 20-valent pneumococcal conjugate vaccine (20vPnC).
  Interventions: Biological: 20-valent pneumococcal conjugate vaccine (20vPnC)

INTERVENTIONS:
Biological: PG4 — Multivalent pneumococcal conjugate vaccine.
  Arms: PG4 1-Dose Group; PG4 2-Dose Group
Biological: 20-valent pneumococcal conjugate vaccine (20vPnC) — 20-valent pneumococcal conjugate vaccine (20vPnC)
  Other Names: Prevnar 20
  Arms: 20-valent pneumococcal conjugate vaccine (20vPnC)

SUMMARY:
The purpose of this study is to learn about the safety, tolerability and immune effects of a pneumococcal vaccine in toddlers.

Participants will take part in this study for approximately 6 or 8 months depending on which group they are assigned to. During this time participants will have 2 clinic visits and 1 phone visit for the 1-Dose group, or 3 clinic visits and 1 phone visit for the 2-Dose group.

At these clinic visits, participants will be asked if any side effects were experienced. The participants will also have to give blood samples during some clinic visits.

ELIGIBILITY:
Inclusion Criteria:

* Male or female toddlers ≥12 to ≤15 months of age at the time of consent.
* Healthy toddlers determined by clinical assessment, including medical history and clinical judgment, to be eligible for the study.
* Have received 3 infant doses of 20vPnC with the last dose administered >56 days before enrollment into the study. Documented confirmation of receipt will be collected prior to randomization.

Exclusion Criteria:

* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis).
* Major known congenital malformation or serious chronic disorder.
* Other acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
* Previous vaccination with any licensed or investigational pneumococcal vaccine (other than 20vPnC) or planned receipt during study participation.

Ages: 12 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 225 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2026-02-16 (Estimated); Study Completion 2026-02-16 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants reporting prespecified local reactions within 7 days after each dose | 7 days after each dose
  Prespecified local reactions (redness, swelling, and pain at the injection site) after each dose
Percentage of participants reporting prespecified systemic events within 7 days after each dose | 7 days after each dose
  Prespecified systemic events (fever, decreased appetite, drowsiness/increased sleep, and irritability) after each dose
Percentage of participants reporting Adverse Events (AEs) within 1 month after the last assigned vaccination | From signing of ICD to 1 month after last assigned vaccination
  Adverse events occurring within 1 month after the last assigned vaccination
Percentage of participants reporting Serious Adverse Events (SAEs) within 6 months after vaccination | From signing of ICD to 6 months after last assigned vaccination
  SAEs occurring from Dose 1 through 6 months after the last assigned vaccination

SECONDARY OUTCOMES:
Pneumococcal serotype specific IgG concentrations | 1 month after last assigned vaccination
  Pneumococcal IgG GMCs 1 month after the last assigned vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (46):
- United States (42):
  - Emerson Clinical Research Institute, Washington D.C., District of Columbia
  - Bio-Medical Research LLC, Miami, Florida
  - Riveldi Biomedical Research and Associates - Miami Lakes, Miami Lakes, Florida
  - Tekton Research, LLC., Chamblee, Georgia
  - Javara - Privia Medical Group Georgia - Fayetteville, Fayetteville, Georgia
  - Rophe Adult and Pediatric Medicine/SKYCRNG, Union City, Georgia
  - Clinical Research Prime, Idaho Falls, Idaho
  - Clinical Research Prime Rexburg, Rexburg, Idaho
  - The Iowa Clinic, Ankeny, Iowa
  - All Children Pediatrics, Louisville, Kentucky
  - Bluegrass Clinical Research, Inc., Louisville, Kentucky
  - Louisiana State University Health Sciences Shreveport - Fairfield avenue, Shreveport, Louisiana
  - Louisiana State University Health Sciences Shreveport, Shreveport, Louisiana
  - Ochsner/LSU Health Ambulatory Care Center, Shreveport, Louisiana
  - University of Maryland, Baltimore, Center for Vaccine Development and Global Health, Baltimore, Maryland
  - University of Maryland, Baltimore, Baltimore, Maryland
  - The Pediatric Center, Columbia, Maryland
  - The Pediatric Center of Frederick, Frederick, Maryland
  - Child Health Care Associates, East Syracuse, New York
  - Atrium Health - Strive Vaccine Research Clinic, Charlotte, North Carolina
  - Atrium Health-Myers Park, Charlotte, North Carolina
  - Duke Vaccine and Trials Unit, Durham, North Carolina
  - Durham Pediatrics at North Duke Street, Durham, North Carolina
  - Atrium Health-Matthews, Matthews, North Carolina
  - Javara - Wake Forest Health Network - Ford, Simpson, Lively & Rice Pediatrics, Winston-Salem, North Carolina
  - Senders Pediatrics, South Euclid, Ohio
  - Cyn3rgy Research, Gresham, Oregon
  - Allegheny Health and Wellness Pavilion, Erie, Pennsylvania
  - Coastal Pediatric Research, Charleston, South Carolina
  - Coastal Pediatric Research, Summerville, South Carolina
  - Holston Medical Group, Kingsport, Tennessee
  - Pediatric Clinical Trials of Tennessee,LLc, Tullahoma, Tennessee
  - Javara - Privia Medical Group North Texas - Dallas, Dallas, Texas
  - Oak Cliff Research Company, LLC, Dallas, Texas
  - PAS Research - McAllen, Edinburg, Texas
  - Mercury Clinical Research - Houston, Houston, Texas
  - DM Clinical Research, Houston, Texas
  - Kool Kids Pediatrics, Houston, Texas
  - Mercury Clinical Research - Sunrise Pediatrics, Houston, Texas
  - Mercury Clinical Research - Pediatric Associates, Houston, Texas
  - University of Texas Medical Branch, League City, Texas
  - Mercury Clinical Research - North Houston Internal Medicine & Pediatric Clinic, Tomball, Texas
- Puerto Rico (4):
  - Ponce Medical School Foundation Inc., Ponce
  - BRCR Medical Center - Ponce, Ponce
  - BRCR Global Puerto Rico, San Juan
  - Caribbean Medical Research Center, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4931010